CLINICAL TRIAL: NCT05018689
Title: Aevidum: Preliminary Evidence to Showcase a Student-Led Mental Health Program
Brief Title: Evaluation of the Aevidum Curriculum and Club
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: The Hollister Confidence Fund (Other)
Responsible Party: Principal Investigator, Deepa Sekhar, Associate Professor, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00017706
Record Dates: First submitted 2021-08-13; First posted 2021-08-24 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Wellness 1
Keywords: Mental Health; Adolescents
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aevidum curriculum (Active Comparator): Curriculum: Aevidum has developed a 5-lesson 3-hour mental health curriculum that can be broken up and integrated into existing school health curricula. The study team in partnership with the Executive Director of Aevidum will collaborate with schools to implement the curriculum to their 9th grade students.
  Interventions: Other: Aevidum curriculum
- Aevidum curriculum + club (Active Comparator): Curriculum + club. Schools assigned to the curriculum plus club will also start an Aevidum club at their school. Club basic processes and ideas for events are housed on the Aevidum website. Schools will select faculty and student leaders who will participate in a kickoff web-based training at the start of the academic year. The training is led by current Aevidum student leaders at schools with successful clubs. This is a standard orientation process that Aevidum has run for many years in-person, but has been adapted to a virtual format with the COVID-19 pandemic.
  Interventions: Other: Aevidum curriculum; Other: Club

INTERVENTIONS:
Other: Aevidum curriculum — The Aevidum curriculum will be delivered to 9th grade students at participating high schools in both study arms. All school staff who plan to deliver the curriculum will participate in a web-based training workshop with the Aevidum Executive Director.
Other: Club — Schools will identify ten students interested in participating in an Aevidum club. Following training of interested students, schools are asked to commit to running two Aevidum club activities during the school year.
  Arms: Aevidum curriculum + club

SUMMARY:
The study purpose is to evaluate the effectiveness of the Aevidum curriculum (plus/minus club) to improve adolescent mental health knowledge, help-seeking intentions, and school culture. Investigators will partner with 12 high schools for this study. Prior to the start of the 2021-2022 academic year, schools will be recruited and randomly assigned to implement the Aevidum curriculum (n=6) or the curriculum and club (n=6). Please note, ultimately a total of 10 schools were recruited, with 5 assigned to each arm.

DETAILED DESCRIPTION:
Aevidum was established in 2009 as a student-led initiative to raise awareness and reduce the stigma surrounding mental illness. Their mental health curriculum and club activities are currently used in over 300 schools in Pennsylvania and surrounding states. In comparison to current interventions, Aevidum is unique in that it provides students the opportunity to build a strong support system among peers. Aevidum's curriculum and club activities provide an opportunity for schools and students to engage with mental health and suicide prevention materials with a student-directed method. Youth voice is a powerful tool that schools and communities can utilize to make mental health and suicide prevention programming more impactful. Allowing youth the chance to lead and let their voices be heard can create greater buy-in for activities.

At present, there is not a strong evidence-base for the efficacy of student-led initiatives that aid in reaching mandated Act 71 curriculum standards for mental health and suicide prevention. Aevidum lacks an evidence-base for its curriculum and club programming, which is freely available to schools. To continue offering free resources, while also maintaining and updating these resources to ensure they are innovative and best reflect student needs, Aevidum needs to establish an evidence-base to support future funding. This project plans to evaluate the effectiveness of these efforts in supporting adolescent mental health. Results will be used to inform school-based mental health programming and to establish an evidence-base for the Aevidum program, furthering mental health awareness and education, while also reducing mental health stigma.

While set up as a randomized clinical trial, this portion of the study is largely exploratory and has not be formally powered. Knowledge, help-seeking, school environment/stigma and program visibility will be assessed both in a pre/post assessment and compared between study arms as follows:

Aim 1: Assess Aevidum's curriculum in improving students' mental health knowledge and help-seeking intentions.

Hypothesis: Exposure to Aevidum's five module mental health curriculum will result in significant improvements in knowledge and help seeking intentions between pre- and post-survey measures using the published University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment among the 6 schools assigned to curriculum only.

Aim 2: Assess the combination of Aevidum's curriculum AND club activities to improve student perceptions of school culture.

Hypothesis: Exposure to both curriculum and club activities will have the added benefit of improving school environment/stigma and program visibility in addition to knowledge and help-seeking on the Peer-to-Peer Depression Awareness Assessment among the 6 schools assigned to curriculum + club.

In secondary statistical analysis, the curriculum-only schools will be compared to the curriculum plus club activities schools directly.

Specifically: 1) Compare students from schools in Aim 1 (curriculum only) to those in Aim 2 (curriculum plus club) regarding changes in knowledge, help-seeking behavior, school environment/stigma and program visibility.

2) Compare the impact on 9th graders in curriculum schools versus 9th graders in curriculum plus club schools (curriculum will specifically be delivered to 9th grade students at all participating high schools).

ELIGIBILITY:
Inclusion Criteria:

* Students (in grades 9-12; this is typically ages 14-18 years though a broader span was provided above) and staff from participating schools.

Exclusion Criteria:

* Students not enrolled in one of the participating high schools (n=12)
* Students not in grades 9-12
* Students with disabilities that are deemed unable to participate by the school district
* Non-English speaking students as curriculum and club materials are taught/available in English only at this time

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2557 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Started | 1560 | 997
Completed | 392 | 345
Not Completed | 1168 | 652

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club | Total
Number analyzed (Participants) | 1560 | 997 | 2557
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.55 (1.22) | 15.71 (1.22) | 15.61 (1.22)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/gender: Male | 764 | 447 | 1211
  Sex/gender: Female | 747 | 515 | 1262
  Sex/gender: Other | 49 | 32 | 81
  Sex/gender: Missing | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic white | 1305 | 886 | 2191
  Race/ethnicity: Non-Hispanic Black | 35 | 13 | 48
  Race/ethnicity: Hispanic | 148 | 51 | 199
  Race/ethnicity: Non-Hispanic Asian | 17 | 21 | 38
  Race/ethnicity: Non-Hispanic Other | 47 | 25 | 72
  Race/ethnicity: Missing | 8 | 1 | 9
Grade [Count of Participants; unit: Participants]
  9th | 506 | 252 | 758
  10th | 398 | 242 | 640
  11th | 369 | 248 | 617
  12th | 279 | 253 | 532
  Missing | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Knowledge Scores From Baseline (1 of 4)
Description: This will be assessed using the University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Response options: 1 Not at all confident, 2-4 Moderately confident, 5-7 Extremely confident
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analyses include p-values from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale
  How confident to identify someone showing depression? | 0.33 [0.21 to 0.45] | 0.29 [0.16 to 0.42]
  How confident to help a friend? | 0.26 [0.11 to 0.42] | 0.24 [0.07 to 0.41]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; How confident to identify someone showing depression?; Test type: Superiority; p = 0.642, Regression, Linear; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.13 to 0.22]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; How confident to help a friend?; Test type: Superiority; p = 0.864, Regression, Linear; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.21 to 0.25]

2. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Knowledge Scores From Baseline (2 of 4)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: If your friend tells you that he/she is thinking about suicide and asks you to keep it a secret because no one else knows, what do you do? Responses are tell someone (correct) or keep it a secret (incorrect).
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analysis includes the p-value from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio | 1.32 [0.94 to 1.84] | 1.70 [1.15 to 2.50]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Test type: Superiority; p = 0.336, Regression, Logistic; comparison of odds ratios = 0.78, 95% CI 2-sided [0.47 to 1.30]

3. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Knowledge Scores From Baseline (3 of 4)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  All responses in this section were true or false. The correct answer (i.e., true or false) to each items is included in the row description below.
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analyses include p-values from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio
  Depression runs in families. Answer: true | 1.41 [1.06 to 1.86] | 1.34 [0.99 to 1.80]
  Depression can be controlled through willpower. Answer: false | 1.31 [1.07 to 1.60] | 1.37 [1.09 to 1.71]
  Depression is treatable. Answer: true | 1.12 [0.86 to 1.46] | 1.21 [0.89 to 1.64]
  Abuse of alcohol and drugs can be a sign of depression. Answer: true | 1.71 [0.98 to 2.97] | 1.54 [0.91 to 2.59]
  Depression is a sign of personal weakness. Answer: false | 1.49 [1.19 to 1.85] | 1.37 [1.03 to 1.82]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Depression runs in families. Answer: true; Test type: Superiority; p = 0.806, Regression, Logistic; comparison of odds ratios = 1.05, 95% CI 2-sided [0.70 to 1.59]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Depression can be controlled through willpower. Answer: false; Test type: Superiority; p = 0.781, Regression, Logistic; comparison of odds ratios = 0.96, 95% CI 2-sided [0.71 to 1.30]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Depression is treatable. Answer: true; Test type: Superiority; p = 0.720, Regression, Logistic; comparison of odds ratios = 0.93, 95% CI 2-sided [0.62 to 1.39]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Abuse of alcohol and drugs can be a sign of depression. Answer: true; Test type: Superiority; p = 0.784, Regression, Logistic; comparison of odds ratios = 1.11, 95% CI 2-sided [0.52 to 2.38]
Statistical Analysis 5: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Depression is a sign of personal weakness. Answer: false; Test type: Superiority; p = 0.662, Regression, Logistic; comparison of odds ratios = 1.08, 95% CI 2-sided [0.76 to 1.55]

4. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Knowledge Scores From Baseline (4 of 4)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  The questions in this section asked students to correctly identify these symptoms of depression (dichotomous responses)
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analyses include p-values from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio
  Difficulty concentrating or making decisions | 1.41 [1.05 to 1.88] | 1.75 [1.24 to 2.47]
  Feeling angry | 1.39 [1.09 to 1.77] | 1.71 [1.30 to 2.25]
  Changes in sleep patterns | 1.38 [0.92 to 2.05] | 1.96 [1.23 to 3.11]
  Frequent unexplained aches and pains | 1.91 [1.57 to 2.34] | 1.71 [1.39 to 2.10]
  Feeling tired or less energetic | 1.88 [1.12 to 3.15] | 0.82 [0.50 to 1.36]
  Eating more than usual | 1.92 [1.52 to 2.43] | 1.90 [1.45 to 2.47]
  Feeling irritable or restless | 1.34 [0.99 to 1.81] | 1.61 [1.12 to 2.32]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Difficulty concentrating or making decisions; Test type: Superiority; p = 0.340, Regression, Logistic; comparison of odds ratios = 0.80, 95% CI 2-sided [0.51 to 1.26]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Feeling angry; Test type: Superiority; p = 0.265, Regression, Logistic; comparison of odds ratios = 0.81, 95% CI 2-sided [0.56 to 1.17]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Changes in sleep patterns; Test type: Superiority; p = 0.259, Regression, Logistic; comparison of odds ratios = 0.70, 95% CI 2-sided [0.38 to 1.30]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Frequent unexplained aches and pains; Test type: Superiority; p = 0.450, Regression, Logistic; comparison of odds ratios = 1.12, 95% CI 2-sided [0.84 to 1.49]
Statistical Analysis 5: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Feeling tired or less energetic; Test type: Superiority; p = 0.025, Regression, Logistic; comparison of odds ratios = 2.28, 95% CI 2-sided [1.11 to 4.69]
Statistical Analysis 6: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Eating more than usual; Test type: Superiority; p = 0.937, Regression, Logistic; comparison of odds ratios = 1.01, 95% CI 2-sided [0.71 to 1.44]
Statistical Analysis 7: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Feeling irritable or restless; Test type: Superiority; p = 0.447, Regression, Logistic; comparison of odds ratios = 0.83, 95% CI 2-sided [0.52 to 1.34]

5. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Help-seeking Intentions Scores From Baseline (1 of 3)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: If you thought that you had depression, how likely is it that you would seek help from the following people or places? Response options: 1 (Not at all likely), 2 (Not too likely), 3 (Somewhat likely), 4 (Very likely)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analyses include p-values from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale
  Friend | 0.05 [-0.03 to 0.13] | 0.03 [-0.06 to 0.12]
  Parent/guardian | 0.0 [-0.08 to 0.09] | 0.05 [-0.04 to 0.15]
  School counselor | 0.13 [0.03 to 0.22] | 0.06 [-0.04 to 0.16]
  Teacher | 0.11 [0.02 to 0.20] | 0.15 [0.05 to 0.24]
  Mental health professional (psychologist, psychiatrist, social worker) | 0.05 [-0.05 to 0.14] | 0.09 [-0.01 to 0.19]
  Doctor | 0.0 [-0.09 to 0.09] | -0.05 [-0.15 to 0.05]
  Internet/website | 0.19 [0.09 to 0.28] | 0.21 [0.11 to 0.31]
  Clergy, priest, rabbi, or other religious person | -0.06 [-0.14 to 0.02] | 0.07 [-0.02 to 0.15]
  Phone helpline | 0.17 [0.08 to 0.25] | 0.11 [0.02 to 0.20]
  Crisis textline | 0.19 [0.10 to 0.27] | 0.11 [0.02 to 0.20]
  Other relative (i.e., sister, brother, aunt, uncle) | -0.03 [-0.13 to 0.06] | 0.02 [-0.08 to 0.12]
  Boyfriend or girlfriend | -0.02 [-0.11 to 0.08] | 0.02 [-0.08 to 0.12]
  Coach | -0.01 [-0.09 to 0.08] | 0.12 [0.02 to 0.21]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Friend; Test type: Superiority; p = 0.800, Regression, Linear; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.11 to 0.14]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Parent/guardian; Test type: Superiority; p = 0.451, Regression, Linear; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.18 to 0.08]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; School counselor; Test type: Superiority; p = 0.335, Regression, Linear; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.07 to 0.2]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Teacher; Test type: Superiority; p = 0.554, Regression, Linear; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.17 to 0.09]
Statistical Analysis 5: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Mental health professional; Test type: Superiority; p = 0.541, Regression, Linear; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.19 to 0.10]
Statistical Analysis 6: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Doctor; Test type: Superiority; p = 0.454, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.09 to 0.19]
Statistical Analysis 7: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Internet/website; Test type: Superiority; p = 0.749, Regression, Linear; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.16 to 0.12]
Statistical Analysis 8: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Clergy, priest, rabbi, or other religious person; Test type: Superiority; p = 0.030, Regression, Linear; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.24 to -0.01]
Statistical Analysis 9: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Phone helpline; Test type: Superiority; p = 0.334, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.06 to 0.18]
Statistical Analysis 10: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Crisis textline; Test type: Superiority; p = 0.243, Regression, Linear; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.05 to 0.20]
Statistical Analysis 11: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Other relative (i.e., sister, brother, aunt, uncle); Test type: Superiority; p = 0.492, Regression, Linear; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.19 to 0.09]
Statistical Analysis 12: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Boyfriend or girlfriend; Test type: Superiority; p = 0.610, Regression, Linear; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.17 to 0.10]
Statistical Analysis 13: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Coach; Test type: Superiority; p = 0.061, Regression, Linear; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.25 to 0.01]

6. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Help-seeking Intentions Scores From Baseline (2 of 3)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Response options yes or no, with preferred answer being "yes" for both items
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analyses include p-values from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio
  If you had depression symptoms for more than 2 weeks, would you ask for help? | 1.10 [0.91 to 1.32] | 0.86 [0.71 to 1.05]
  If you thought you had mental health issues, is there a trusted adult you would go to? | 1.28 [0.99 to 1.67] | 1.14 [0.86 to 1.50]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; If you had depression symptoms for more than 2 weeks, would you ask for help?; Test type: Superiority; p = 0.086, Regression, Logistic; comparison of odds ratios = 1.27, 95% CI 2-sided [0.97 to 1.66]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; If you thought you had mental health issues, is there a trusted adult you would go to?; Test type: Superiority; p = 0.526, Regression, Logistic; comparison of odds ratios = 1.13, 95% CI 2-sided [0.77 to 1.66]

7. Primary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Help-seeking Intentions Scores From Baseline (3 of 3)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: Do you know how to get help in your school? Response options: 1 (Not really), 2 (Sort of), 3 (Definitely)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analysis includes the p-value from a mixed effects linear regression model.
Time Frame: baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale | 0.11 [0.05 to 0.17] | 0.05 [-0.02 to 0.12]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Do you know how to get help in your school?; Test type: Superiority; p = 0.199, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.03 to 0.16]

8. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (1 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: Imagine that you recently heard about a new student at your school who has depression. To what extent do you agree or disagree with the following statements? Response options: 1 (strongly disagree), 2 (disagree), 3 (neither agree nor disagree), 4 (agree), 5 (strongly agree)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analyses include p-values from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale
  The new student is more dangerous than other students | -0.10 [-0.19 to -0.01] | 0.15 [0.05 to 0.25]
  The student is to blame for his or her condition | -0.11 [-0.19 to -0.03] | 0.07 [-0.02 to 0.15]
  I would have sympathy for the new student | -0.02 [-0.10 to 0.06] | -0.08 [-0.16 to 0.01]
  The new student makes me feel scared | -0.02 [-0.10 to 0.06] | 0.07 [-0.01 to 0.16]
  The new student makes me feel uncomfortable | 0.03 [-0.05 to 0.12] | 0.01 [-0.08 to 0.10]
  I would help the new student even if I did not know him or her well | -0.09 [-0.17 to -0.01] | -0.21 [-0.30 to -0.13]
  I would try to stay away from the new student | -0.06 [-0.14 to 0.03] | 0.12 [0.03 to 0.21]
  The new student would be made fun of at my school | 0.17 [0.08 to 0.26] | 0.19 [0.09 to 0.29]
  The new student would be ignored at my school | 0.08 [-0.01 to 0.17] | 0.17 [0.07 to 0.27]
  I think other students in my school would try to help the new student | -0.13 [-0.22 to -0.04] | -0.16 [-0.26 to -0.06]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The new student is more dangerous than other students; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.38 to -0.12]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The student is to blame for his or her condition; Test type: Superiority; p = 0.003, Regression, Linear; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.29 to -0.06]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; I would have sympathy for the new student; Test type: Superiority; p = 0.310, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.06 to 0.18]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The new student makes me feel scared; Test type: Superiority; p = 0.114, Regression, Linear; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.21 to 0.02]
Statistical Analysis 5: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The new student makes me feel uncomfortable; Test type: Superiority; p = 0.738, Regression, Linear; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.10 to 0.15]
Statistical Analysis 6: Comparison: Aevidum Curriculum; I would help the new student even if I did not know him or her well; Test type: Superiority; p = 0.040, Regression, Linear; Mean Difference (Net) = 0.12, 95% CI 2-sided [0.01 to 0.24]
Statistical Analysis 7: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; I would try to stay away from the new student; Test type: Superiority; p = 0.006, Regression, Linear; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.29 to -0.05]
Statistical Analysis 8: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The new student would be made fun of at my school; Test type: Superiority; p = 0.798, Regression, Linear; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.15 to 0.11]
Statistical Analysis 9: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; The new student would be ignored at my school; Test type: Superiority; p = 0.197, Regression, Linear; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.22 to 0.05]
Statistical Analysis 10: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; I think other students in my school would try to help the new student; Test type: Superiority; p = 0.623, Regression, Linear; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.10 to 0.16]

9. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (2 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: On a scale from 1 to 7, if you were seen going into the office of your school social worker or school psychologist, how would you feel? Response options: 1 (Not at all embarrassed), 2, 3, 4 (Moderately embarrassed), 5, 6, 7 (Extremely embarrassed)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analysis includes the p-value from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale | -0.16 [-0.33 to 0.02] | -0.21 [-0.39 to -0.02]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; On a scale from 1 to 7, if you were seen going into the office of your school social worker or school psychologist, how would you feel?; Test type: Superiority; p = 0.718, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.21 to 0.30]

10. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (3 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: How comfortable are you talking about mental health issues with other students at your school? Response options: 1 (Not at all comfortable), 2, 3, 4 (Moderately comfortable), 5, 6, 7 (Extremely comfortable)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analysis includes the p-value from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale | 0.36 [0.19 to 0.53] | 0.15 [-0.04 to 0.33]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; How comfortable are you talking about mental health issues with other students at your school?; Test type: Superiority; p = 0.090, Regression, Linear; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.03 to 0.46]

11. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (4 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: What mental health issues do you think are most concerning to other students at your school? Response options: dichotomous response for each listed mental health issue in rows below
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analyses include p-values from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio
  Depression | 0.98 [0.76 to 1.28] | 1.00 [0.76 to 1.32]
  Anxiety | 1.22 [0.94 to 1.57] | 1.03 [0.81 to 1.33]
  Thoughts of suicide | 1.18 [0.95 to 1.46] | 1.10 [0.85 to 1.41]
  I do not think there are any mental health issues that are concerning for students | 1.01 [0.67 to 1.53] | 1.28 [0.84 to 1.94]
  Other | 4.24 [3.16 to 5.68] | 4.87 [3.51 to 6.77]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Depression; Test type: Superiority; p = 0.944, Regression, Logistic; comparison of odds ratios = 0.99, 95% CI 2-sided [0.67 to 1.44]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Anxiety; Test type: Superiority; p = 0.369, Regression, Logistic; comparison of odds ratios = 1.18, 95% CI 2-sided [0.82 to 1.68]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Thoughts of suicide; Test type: Superiority; p = 0.676, Regression, Logistic; comparison of odds ratios = 1.07, 95% CI 2-sided [0.77 to 1.50]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; I do not think there are any mental health issues that are concerning for students; Test type: Superiority; p = 0.432, Regression, Logistic; comparison of odds ratios = 0.79, 95% CI 2-sided [0.44 to 1.42]
Statistical Analysis 5: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Other; Test type: Superiority; p = 0.533, Regression, Logistic; comparison of odds ratios = 0.87, 95% CI 2-sided [0.56 to 1.35]

12. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (5 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Response options: 1 (A little), 2 (some), 3 (A lot)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analyses include p-values from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale
  How much do your teachers know about addressing student mental health needs? | 0.0 [-0.06 to 0.07] | 0.02 [-0.05 to 0.09]
  How much do your school counselors know about addressing student mental health needs? | 0.04 [-0.03 to 0.11] | -0.02 [-0.09 to 0.06]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; How much do your teachers know about addressing student mental health needs?; Test type: Superiority; p = 0.769, Regression, Linear; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.11 to 0.08]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; How much do your school counselors know about addressing student mental health needs?; Test type: Superiority; p = 0.315, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.05 to 0.16]

13. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (6 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: How would you like your school to show that they care about student mental health? Response options: dichotomous for each item listed below
  Results provided in the outcome measure data table include odds of a correct response from pre to post test reported in each study arm as odds ratio (95% CI). Statistical analyses include p-values from a mixed effects logistic regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
odds ratio
  Mental health information sheets at school | 0.86 [0.70 to 1.06] | 1.0 [0.79 to 1.26]
  Class activities about mental health | 0.86 [0.71 to 1.05] | 0.88 [0.70 to 1.10]
  Mental health information on school website | 0.97 [0.78 to 1.20] | 0.89 [0.71 to 1.12]
  Other | 3.84 [3.01 to 4.89] | 3.36 [2.55 to 4.42]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Mental health information sheets at school; Test type: Superiority; p = 0.345, Regression, Logistic; comparison of odds ratios = 0.86, 95% CI 2-sided [0.63 to 1.18]
Statistical Analysis 2: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Class activities about mental health; Test type: Superiority; p = 0.899, Regression, Logistic; comparison of odds ratios = 0.98, 95% CI 2-sided [0.73 to 1.33]
Statistical Analysis 3: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Mental health information on school website; Test type: Superiority; p = 0.612, Regression, Logistic; comparison of odds ratios = 1.08, 95% CI 2-sided [0.80 to 1.48]
Statistical Analysis 4: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Other; Test type: Superiority; p = 0.476, Regression, Logistic; comparison of odds ratios = 1.14, 95% CI 2-sided [0.79 to 1.65]

14. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (7 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: On average, how often do your teachers speak to you about your emotions and feelings? Response options: 1 (daily), 2 (weekly), 3 (monthly), 4 (never)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analysis includes the p-value from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale | -0.08 [-0.16 to 0.0] | 0.01 [-0.08 to 0.10]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; On average, how often do your teachers speak to you about your emotions and feelings?; Test type: Superiority; p = 0.141, Regression, Linear; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.22 to 0.03]

15. Secondary Outcome: Change in University of Michigan Depression Center Peer-to-Peer Depression Awareness Assessment Perceptions of School Culture Scores From Baseline (8 of 8)
Description: This will be assessed using the University of Michigan Depression Center (UMDC) Peer-to-Peer Depression Awareness Assessment:
  baseline assessment (pre-intervention) at the start of the school year and post-assessment after curriculum +/- club delivery (an average of 9 months)
  Question: Would you like your teachers to speak to you about your emotions and feelings? Response options: 1 (yes), 2 (maybe), 3 (no)
  Results provided in the outcome measure data table include difference of mean score from pre to post test (95% CI) in each study arm. Statistical analysis includes the p-value from a mixed effects linear regression model.
Time Frame: baseline (pre-intervention) and post-study completion (an average of 9 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
Number analyzed (Participants) | 1560 | 997
score on a scale | 0.0 [-0.07 to 0.06] | -0.04 [-0.11 to 0.02]
Statistical Analysis 1: Comparison: Aevidum Curriculum vs Aevidum Curriculum + Club; Would you like your teachers to speak to you about your emotions and feelings?; Test type: Superiority; p = 0.392, Regression, Linear; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.05 to 0.13]

ADVERSE EVENTS:
Description: As this was an educational curriculum and club evaluation, all-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Aevidum Curriculum | Aevidum Curriculum + Club
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05018689/Prot_SAP_000.pdf